CLINICAL TRIAL: NCT04261023
Title: Phase II Proof of Concept Study of Abatacept (Orencia) in Individuals Who aRe Considered At Risk of Developing Inflammatory Arthritis
Brief Title: Abatacept in Individuals Who aRe Considered At Risk of Developing Inflammatory Arthritis
Acronym: ARCADIA
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: The CI terminated ARCADIA early due to a number of reasons. These include the difficulty in recruiting and being placed on pause during the COVID pandemic, plus limited staffing at that time & the need to considerably amend the eCRF MACRO system
Sponsor: University of Leeds (Other)
Responsible Party: Principal Investigator, Paul Emery, Professor of Rheumatology, University of Leeds
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: RR15/348
Record Dates: First submitted 2020-01-30; First posted 2020-02-07 (Actual); Last update posted 2025-03-30 (Actual); Status verified 2025-03

CONDITIONS: Inflammatory Arthritis
Keywords: Abatacept (Orencia)
MeSH Terms: conditions — Arthritis | interventions — Abatacept

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Abatacept (Experimental): Treatment arm - 125mg sub-cutaneous injection at week 0 and once weekly thereafter for a maximum of 48 weeks
  Interventions: Drug: Orencia 125 MG Per 1 ML Prefilled Syringe
- Control arm - CCP Next Generation (No Intervention): Observational study cohort - usual care

INTERVENTIONS:
Drug: Orencia 125 MG Per 1 ML Prefilled Syringe — Abatacept sub-cutaneous injection 125mg at week 0 and once weekly thereafter for a maximum of 48 weeks
  Other Names: Abatacept
  Arms: Abatacept

SUMMARY:
Phase II, single-centre, open label, two parallel arm cohort randomised controlled trial (RCT) testing abatacept in a population of anti-CCP Ab positive individuals at moderate to high risk of developing IA according to a published risk score, already followed in the observational study 'CCP: Next Generation'

DETAILED DESCRIPTION:
There is now evidence that the immunological disease process starts many years before the onset of clinically detectable inflammatory arthritis (IA). It is now a realistic goal to treat individuals in this pre-clinical phase with the possibility of arresting their progression to clinical disease.

Individuals at risk of developing RA can be identified by the presence of CCP antibodies alongside other clinical features. In Leeds we have developed a prediction model that stratifies these individuals into at-risk vs. low risk. At present there are no treatments in this pathway until individuals develop IA.

T-cells appear to be an appropriate target in at-risk individuals as they play a critical role in the generation and maintenance of autoimmunity. Abatacept (Orencia) is a selective T-cell modulator that blocks a co-stimulatory signal needed to activate T-cells and has an excellent safety profile.

ELIGIBILITY:
Inclusion Criteria:

* Participant in Leeds CCP 'Next Generation' observational cohort who has tested positive for anti-CCP Ab and accepted to be approached for a interventional study
* Age >18 years old.
* At moderate to high risk of progression to IA (see below).
* Consents to be contacted in future for an interventional study

A prediction model will be used to risk stratify individuals based on the following predictors:

1. Tenderness of ≥1 small joint of the hands or feet defined by the physician (one point)
2. Early morning stiffness ≥30 minutes (one point)
3. RF and/or anti-CCP Ab concentration >3x upper limit of normal. (2 points) The participant's risk will be calculated according to the model suggested by Rakieh et al. (1). Those with a score of ≥3 out of 4 will be eligible to be randomised.

   * For the intervention arm:

     * Randomised to intervention arm
     * Consents to commence Abatacept therapy (if not, will remain in CCP Next-generation study)
   * For the control arm:

     * Randomised to the control arm
     * Will remain in the CCP Next-generation study

Exclusion Criteria:

For both the intervention and control arms:

* Previous diagnosis of RA or other form of inflammatory arthritis including, but not limited to SLE, psoriatic arthritis, ankylosing spondylitis, gout or pyrophosphate arthropathy and including current treatment with DMARDs or biological therapy
* Clinical synovitis on clinical examination by a rheumatologist
* Presence of concomitant illness likely to require systemic glucocorticosteroid therapy during the study, in the opinion of the investigator
* Treatment with an intravenous, intramuscular, intrabursal or intraarticular corticosteroid within 12 weeks prior to randomization
* Co-morbidities requiring chronic treatment with immunosuppressive or immune modulating therapy.
* Women in the intervention arm who get pregnant during the study will be withdrawn from treatment and followed for the duration of the pregnancy for safety purposes. All participants who get pregnant will continue to be followed up in clinic as standard NHS care to collect secondary end point data
* Evidence of active or latent bacterial or viral infection at the time of potential enrolment, including human immunodeficiency or herpes zoster virus or cytomegalovirus that resolved less than 2 months prior to enrolment
* Individuals with palindromic rheumatism

For the intervention arm only:

* History of acute allergic reactions to biologic therapies or immunoglobulins
* Subjects with current symptoms of severe, progressive, or uncontrolled renal, hepatic, hematologic, gastrointestinal, pulmonary, cardiac, neurologic, or cerebral disease, whether or not related to RA and which, in the opinion of the investigator, might place a subject at unacceptable risk for participation in the study
* Subjects who have at any time received treatment with any investigational drug within 28 days of the first dose of study drug
* Subjects who test positive for Hepatitis B, C or HIV.
* Subjects with tuberculosis (TB), including those at high risk of TB, chronic viral infections, recent serious bacterial infections, subjects receiving live vaccinations within 3 months of the anticipated first dose of study medication, or those with chronic illnesses that would, in the opinion of the investigator, put the participant at risk
* Subjects who currently abuse drugs or alcohol
* Subjects with a history of cancer in the last 5 years, other than non-melanoma skin cell cancers cured by local resection or carcinoma in situ
* Scheduled for or anticipating joint replacement surgery
* Men or women unwilling to use an acceptable method of contraception (detailed in 7.1.4) to avoid pregnancy for up to 14 weeks after the last dose of trial medication
* Women of childbearing potential with a positive serum or urine pregnancy test within 48 hours prior to the baseline visit. Women of child bearing potential are defined as women who have had any menstrual bleeding in the last 24 months and who have not had a hysterectomy or surgical sterilisation
* Evidence of active or latent bacterial or viral infection at the time of potential enrolment, including human immunodeficiency or herpes zoster virus or cytomegalovirus that resolved less than 2 months prior to enrolment
* Inadequate haematological, hepatic or renal function within 28 days of treatment:

  * Haemoglobin <8.5 g/dL
  * White blood cells <3000/mm3
  * Platelets <100,000/mm3
  * Serum creatinine, ALT or AST >2 times upper limit of normal
  * Any other laboratory test result that, in the opinion of the study investigator, might place the participant at unacceptable risk for participation in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2020-02-24 (Actual); Primary Completion 2021-03-15 (Actual); Study Completion 2021-03-15 (Actual)

PRIMARY OUTCOMES:
Individuals who develop inflammatory arthritis | 48 weeks
  The percentage of individuals that have developed inflammatory arthritis at 48 weeks

SECONDARY OUTCOMES:
Acute phase reactant levels | Weeks 12, 24, 36, 48, 60, 72, 84 and 96
  Acute phase reactant levels at weeks 12, 24, 36, 48, 60, 72, 84 and 96
Ultrasound synovitis and erosions | Weeks 24, 48, 72 and 96
  Power Doppler to record quantitative scoring 0-3 and erosions
Plain radiograph | Weeks 48 and 96
  Plain radiograph Sharp Van der Heide score 0-5
Patient-reported measures | Weeks 12, 24, 36, 48, 60, 72, 84 and 96
  Physician assessment of global disease activity 0-100mm
Joint swelling and tenderness | Weeks 12, 24, 36, 48, 60, 72, 84 and 96
  28/44 joint count of all tender and swollen joints via diagram
T-cell subset levels | Weeks 12, 24, 36, 48, 60, 72, 84 and 96
  T-cell subset levels
Toxicity levels | Weeks 12, 24, 36, 48, 60, 72, 84 and 96
  Toxicity levels according to the common toxicity criteria gradings

CONTACTS AND LOCATIONS:
Locations (1):
- Institute of Rheumatic & Musculoskeletal Medicine, Chapel Allerton Hospital, Leeds, WEST Yorkshire, United Kingdom